CLINICAL TRIAL: NCT04324190
Title: Online Support for Psychosocial Stress in the Context of the COVID-19 Pandemic
Brief Title: DIgital Online SuPport for COVID-19 StrEss
Acronym: DISPOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gunther Meinlschmidt (Other)
Collaborators: Selfapy GmbH (Unknown)
Responsible Party: Sponsor-Investigator, Gunther Meinlschmidt, Prof. Dr., International Psychoanalytic University Berlin
Organization: International Psychoanalytic University Berlin (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IPUB_2020_01
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Psychosocial Stress; Mental Health
Keywords: COVID-19; SARS-CoV-2; psychosocial stress; online support; guided; mental health; anxiety; depression; somatic symptom disorder
MeSH Terms: conditions — COVID-19; Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with a waiting comparator condition (provision of WHO recommendations, comparable to treatment as usual, TAU), consisting of a two weeks waiting period during which general WHO recommendations how to handle stress in the context of the COVID-19 pandemic will be provided. All subjects in the waiting condition will undergo the intervention following the waiting period. Main assessments will be conducted before the waiting period, before beginning of the intervention, two weeks after beginning of the intervention (+2 weeks), +4 weeks, +12 weeks, and follow ups at +6 months and +12 months.
Who Masked: Care Provider
Masking Description: Care providers (providing guidance) are not informed about wether participants have been assigned to the online support program condition or the comparator condition, consisting of a waiting period followed by the online support program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online support program (Experimental): Guided online support program, consisting of modules (structured in chapters) aiming at reduce stress related to the COVID-19 pandemic.
  Interventions: Behavioral: Guided online support program
- Waiting period (WHO recommendation) (Active Comparator): Waiting period (2 weeks duration) during which subjects are provided with the WHO recommendations "Coping with stress during the 2019 nCoV outbreak". Following the 2 weeks waiting period, subjects are provided with the guided online support program outlined in the arm 'online support program'.
  Interventions: Behavioral: Guided online support program; Behavioral: WHO recommendations (waiting condition)
- No intervention (natural course) (No Intervention): This non-randomised arm (recruited separately; anticipated sample size of 500 subjects, not counted in the overall anticipated sample size) consists of subjects not intending to participate in the Selfapy online support program. Assessment points in this arm are comparable to those in the arm "Online support program" (in the 'No intervention (natural course)' arm, T1 refers to time of study inclusion).

INTERVENTIONS:
Behavioral: Guided online support program — Guided online support program consisting of several modules; Module "General information ..." is an unspecific control module (providing general information on hygiene etc. with no expected effect on outcomes)
  Other Names: online intervention; guided online support
  Arms: Online support program; Waiting period (WHO recommendation)
Behavioral: WHO recommendations (waiting condition) — During the waiting period, a german translation of the WHO recommendations "Coping with stress during the 2019-nCoV outbreak" is provided
  Arms: Waiting period (WHO recommendation)

SUMMARY:
The COVID-19 pandemic leads to a greatly increased risk of substantial psychological stress worldwide. We intend to evaluate an online support program aiming at reducing stress in the context of the COVID-19 pandemic. The program consists of twelve modules that participants undergo, covering a broad range of topics related to stress in the context of the COVID-19 pandemic. It has been developed together with and is provided by Selfapy GmbH, Berlin. The aim of this randomised clinical trial with observational components is to estimate the effects of the intervention as a whole, as well as individual modules and selected chapters. Further, follow-up assessments as well as information on risks and the long-term course of COVID pandemic-related stress may help to elucidate COVID-19 pandemic stress across time and what we can do to prevent long-term negative consequences.

DETAILED DESCRIPTION:
The overall aim of this randomised trial with observational component is to estimate the effects of a guided digital online support program to increase mental health and reduce psychosocial stress in the context of the COVID-19 pandemic. More specifically, the main hypothesis is to estimate whether the improvement in mental health is stronger during the first two weeks of applying the online support program as compared to a two weeks waiting condition (with provision of WHO information on 'coping with stress during the 2019-nCoV' outbreak only). In addition to the randomised control group (second arm: waiting condition, followed by online support program), the study comprises as third arm a non-randomised comparator condition, consisting of subjects not intending to participate in the online support program. Furthermore, our aim is to estimate changes in the outcomes along taking part in the program.

Additional research questions are:

* to compare the intervention effects across modules and chapters of the online support program, including between module comparison with an unspecific, control (comparator) module: "general information on the corona virus" and its unspecific chapters;
* to estimate the effects of selected modules on additional outcomes (e.g. physical activity, and schooling related factors);
* to describe the magnitude and course of psychosocial stress, mental health and related factors in the context of the COVID-19 pandemic;
* to estimate and predict which subjects profit most from specific parts of the program.

Follow-up assessment shall include estimating whether the program prevents the development of detrimental mental health conditions, e.g. depression, anxiety, etc.

In order to make first study results available as early as possible, we intend to conduct quick complete analyses (primary outcome and relevant parts of secondary/other outcomes): These analyses will be conducted with data including subjects from the first 4 weeks of recruitment, given that a sample size of at least 300 for the online support program arm and a sample size of at least 300 for the waiting condition is reached; or if not yet reached after 4 weeks of recruitment, as soon as a sample size of at least 300 for the online support program arm and a sample size of at least 300 for the waiting condition is reached. However, we intend to continue recruiting beyond this point in time and sample size (until the COVID-19 pandemic situation has come to an end, i.e., vaccination is broadly available), to allow further, also more detailed analyses at a later point in time, resulting in more precise estimates.

ELIGIBILITY:
Inclusion criteria, general:

* Sufficient German language skills to participate in the assessments.
* Providing informed consent for participation.

Inclusion criteria for the arms "Online support program" and "Waiting condition...":

- Having signed up for the online support program provided by selfapy GmbH, Berlin, Germany (www.selfapy.de/corona) aiming at reducing burden in the context of the COVID-19 pandemic.

Inclusion criteria for the arm "No intervention...":

- Not having signed up for the online support program provided by selfapy GmbH, Berlin, Germany (www.selfapy.de/corona) aiming at reducing burden in the context of the COVID-19 pandemic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Short-Form-36 (SF-36) Health Survey - Mental Health Component Summary score | Change from T1 (baseline before online support - day 1) to T2 (T1 + 2 weeks) in arm 1, versus change from T0 (baseline before waiting) to T1 (baseline before online support) in arm 2
  The SF-36 is a widely used patient-reported outcome assessment tool to measure health-related quality of life and has high acceptability. The SF-36 is a standardised questionnaire with good psychometric properties.

SECONDARY OUTCOMES:
Short-Form-36 (SF-36) Health Survey - Mental Health Component Summary score | T2 (T1+2 weeks) (arm 2 only), T3 (T1+4 weeks), T4 (T1+12 weeks), follow ups: T1+ 6 months, T1+12 months
  mental health related quality of life
Chronic stress items (9 items) | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T2 (T1+2 weeks), T3 (T1+4 weeks), T4 (T1+12 weeks), follow ups: T1+ 6 months, T1+12 months
  Assessing chronic stress (Petrowski et al., 2019)
Generalized Anxiety Disorder Scale (GAD-7) | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T2 (T1+2 weeks), T3 (T1+4 weeks), T4 (T1+12 weeks), follow ups: T1+ 6 months, T1+12 months
  Assessing anxiety symptoms (Löwe et al., 2008)
Patient Health Questionnaire (PHQ8) | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T2 (T1+2 weeks), T3 (T1+4 weeks), T4 (T1+12 weeks), follow ups: T1+ 6 months, T1+12 months
  Assessing depressive symptoms (Kroenke et al., 2001)
Somatic Symptom Disorder (SSD-12) | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T2 (T1+2 weeks), T3 (T1+4 weeks), T4 (T1+12 weeks), follow ups: T1+ 6 months, T1+12 months
  Assessing depressive symptoms (Toussaint et al., 2019)
Somatic Symptom Scale (SSS-8) | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T2 (T1+2 weeks), T3 (T1+4 weeks), T4 (T1+12 weeks), follow ups: T1+ 6 months, T1+12 months
  Assessing somatic symptoms (Gierk et al., 2015)
Allgemeine Selbstwirksamkeit Kurzskala (ASKU) | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T2 (T1+2 weeks), T3 (T1+4 weeks), T4 (T1+12 weeks), follow ups: T1+ 6 months, T1+12 months
  competence expectations to deal with difficulties and obstacles in daily life (Beierlein et al., 2014)
Screening Tool for Psychological Distress (STOP-D) - selected items | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T1+2 weeks, T1+4 weeks, T1+12 weeks, follow ups: T1+ 6 months, T1+12 months; before & after each module of the online intervention
  stress, anxiety, depression, social support - single item assessments to be applied repeatedly along the online support intervention (Young, Ignaszewski, Fofonoff, Kaan; 2007), including stress of children and anticipation

OTHER OUTCOMES:
Physical activity | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T1+2 weeks, T1+4 weeks, T1+12 weeks, follow ups: T1+ 6 months, T1+12 months; before & after sports and physical activity module; at baseline: before COVID-19 pandemic
  Vigorous, moderate, and walking activity (minutes/day)
Home-schooling | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T1+2 weeks, T1+4 weeks, T1+12 weeks, follow ups: T1+ 6 months, T1+12 months; before & after sports and physical activity module; at baseline: before COVID-19 pandemic
  Questions related to home-schooling related stress & learning
Information related to COVID-19 and SARS-CoV-2 | baseline before waiting (T0, arm 2 only); baseline before online support (day 1, T1), T1+2 weeks, T1+4 weeks, T1+12 weeks, follow ups: T1+ 6 months, T1+12 months; before & after the sports and physical activity module of the online intervention
  Questions related to COVID-19 and SARS-CoV-2 symptoms, disease, and testing, anxiety, stressors
Unintended effects | only after undergoing online support program: T1+2 weeks, T1+4 weeks, T1+12 weeks, follow ups: T1+ 6 months, T1+12 months
  Unintended effects of online support program

CONTACTS AND LOCATIONS:
Locations (1):
- Selfapy GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No